CLINICAL TRIAL: NCT02224664
Title: A Phase 1b, 2-period, Open Label, Multicenter, Dose Escalation Study To Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Pf-06649751 In Subjects With Parkinson's Disease And Motor Fluctuations
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of PF-06649751 in Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Basic Science
Other Study IDs: B7601005; 2014-003472-22 (EudraCT Number)
Record Dates: First submitted 2014-08-15; First posted 2014-08-25 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2016-12

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 3 (Experimental): Titration of PF-06649751 up to 5 mg QD
  Interventions: Drug: PF-06649751
- Cohort 4 (Experimental): Titration of PF-06649751 up to 15 mg QD
  Interventions: Drug: PF-06649751
- Cohort 5 (Experimental): Titration of PF-06649751 up to 15 mg QDi n subjects with Levodopa-induced dyskinesias (LID)
  Interventions: Drug: PF-06649751
- Cohort 6 (Experimental): Titration of PF-0649751 up to 25 mg QD
  Interventions: Drug: PF-06649751

INTERVENTIONS:
Drug: PF-06649751 — Oral daily doses titrated up to 5mg QD
  Arms: Cohort 3
Drug: PF-06649751 — Oral daily doses titrated up to 15 mg QD
  Arms: Cohort 4
Drug: PF-06649751 — Oral daily doses titrated up to 15 mg QD (slow titration with option to down titrate)
  Arms: Cohort 5
Drug: PF-06649751 — Oral daily doses titrated up to 25 mg QD
  Arms: Cohort 6

SUMMARY:
This study will be an open label, dose escalation study to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of repeated daily quaque die (QD) doses given over 21 days (Day 3 to Day 23) to sequential cohorts of subjects with Parkinson's disease. Each cohort will have 2 study periods. For each cohort, subjects will enter Period 1 and if they meet criteria, approximately 12 subjects will be enrolled into Period 2 and dosed with PF 06649751. Based on results observed in a previous study, Cohorts 1 and 2 will not be conducted. Cohorts 3 - 6 will test doses uptitrated to 5 mg, 15 mg and 25 mg QD. Doses may be modified based on emerging safety, tolerability and PK data, but the maximum daily dose that will be given in any cohort will have PK predictions at steady state that are anticipated to be below toxicokinetic limits. An option for down titration to the previous dose level is available should the investigator consider that an AE is intolerable. Following down titration, a single up titration to the next dose level may be attempted if the subject remains symptom free for at least 48 hrs. Safety, tolerability and PK data of Cohort 3 will be reviewed prior to initiating the dosing in Cohorts 4 and 5. Available safety, tolerability and PK data up to Day 24 of at least 5 subjects from Cohorts 4 will be reviewed prior to initiating the dosing in Cohort 6.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic Parkinson's Disease with at least 2 out of 3 cardinal characteristics (tremor, rigidity, bradykinesia)
* Mini-Mental State Examination (MMSE) ≥ 25
* Hoehn & Yahr Stage I-III inclusive
* Documented history of end of L-Dopa wearing OFF
* Cohort 5 only: History of dyskinesia following L-Dopa dosing and Score of at least 2 on Part IV, item 4.2 (functional impact of dyskinesia) of the MDS-UPDRS

Exclusion Criteria:

* Atypical/secondary parkinsonism
* History of surgical intervention for Parkinson's Disease
* Dementia/cognitive impairment that can interfere with study assessments

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- United States (16):
  - Orange Coast Memorial Medical Center, Fountain Valley, California
  - The Parkinson's and Movement Disorder Institute, Fountain Valley, California
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - Rocky Mountain Movement Disorders Center, Englewood, Colorado
  - Davita Clinical Research Center, Lakewood, Colorado
  - MD Clinical, Hallandale, Florida
  - Compass Research, LLC, Orlando, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Massachusetts General Hospital -- FOR DRUG SHIPMENT ONLY, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Quest Research Institute, Farmington Hills, Michigan
  - PRA International, Marlton, New Jersey
  - Carolina Phase I Research, LLC, Raleigh, North Carolina
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Neurology Consultants of Dallas, PA, Dallas, Texas
  - Walnut Hill Medical Center, Dallas, Texas
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- [Derived] Sohur US, Gray DL, Duvvuri S, Zhang Y, Thayer K, Feng G. Phase 1 Parkinson's Disease Studies Show the Dopamine D1/D5 Agonist PF-06649751 is Safe and Well Tolerated. Neurol Ther. 2018 Dec;7(2):307-319. doi: 10.1007/s40120-018-0114-z. Epub 2018 Oct 25. PMID 30361858
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7601005&StudyName=Safety%2C%20Tolerability%2C%20Pharmacokinetics%20and%20Pharmacodynamics%20of%20PF-06649751%20in%20Parkinson%60s%20Disease%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study consists of 2 periods: Lead-in period (Period 1) and dose escalation period (Period 2). Participants were enrolled in Lead-in period only. Participants completed the lead-in period entered into dose escalation period.
Groups:
- L-Dopa: Participants received a single oral tablet/capsule of L-Dopa on Day 1 of first intervention period. Dose ranges from 50 milligram (mg) up to a maximum dose of 250 mg, based on investigator's discretion in Period 1.
- PF-06649751 5 mg + L-Dopa: Participants received a single oral tablet of PF-06649751 once daily along with L-Dopa oral tablets (dose of L-Dopa was based on investigator's decision) from Day 3 up to Day 23 in Period 2. Dose levels were titrated from 0.25 mg up to a maximum dose level of 5 mg.
- PF-06649751 15 mg + L-Dopa: Participants received a single oral tablet of PF-06649751 once daily along with L-Dopa oral tablets (dose of L-Dopa was based on investigator's decision) from Day 3 up to Day 23 in Period 2. Dose levels were titrated from 1.0 mg up to a maximum dose of 15 mg.
- PF-06649751 15 mg + L-Dopa: L-dopa Induced Dyskinesia (LID): Participants with LID received a single oral tablet of PF-06649751 once daily along with L-Dopa oral tablets (dose of L-Dopa was based on investigator's decision) from Day 3 up to Day 23 in Period 2. Dose levels were titrated from 1 mg up to a maximum dose level of 15 mg.
- PF-06649751 25 mg + L-Dopa: Participants received a single oral tablet of PF-06649751 once daily along with L-Dopa oral tablets (dose of L-Dopa was based on investigator's decision) from Day 3 up to Day 23 in Period 2. Dose levels were titrated from 1 mg up to a maximum dose level of 25 mg.
Period: Lead-in Period (3 Days)
Arm/Group | L-Dopa | PF-06649751 5 mg + L-Dopa | PF-06649751 15 mg + L-Dopa | PF-06649751 15 mg + L-Dopa: L-dopa Induced Dyskinesia (LID) | PF-06649751 25 mg + L-Dopa
Started | 50 | 0 | 0 | 0 | 0
Completed | 45 | 0 | 0 | 0 | 0
Not Completed | 5 | 0 | 0 | 0 | 0
Not completed — Does not meet entrance criteria | 5 | 0 | 0 | 0 | 0
Period: Dose Escalation Period (21 Days)
Arm/Group | L-Dopa | PF-06649751 5 mg + L-Dopa | PF-06649751 15 mg + L-Dopa | PF-06649751 15 mg + L-Dopa: L-dopa Induced Dyskinesia (LID) | PF-06649751 25 mg + L-Dopa
Started | 0 | 9 | 11 | 6 | 19
Completed | 0 | 9 | 9 | 3 | 8
Not Completed | 0 | 0 | 2 | 3 | 11
Not completed — Adverse Event | 0 | 0 | 2 | 2 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 4

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who received at least 1 dose of study medication (L-Dopa or PF-06649751) in Period 1 and/or Period 2.
Groups:
- Overall Study: All participants who received a single oral dose of L-Dopa tablet/capsule (up to a maximum dose of 250 mg, based on investigator's discretion) in lead-in period and/or single oral dose of PF-06649751 tablet (3 mg, 5 mg, 15 mg and 25 mg) in dose escalation period.
Arm/Group | Overall Study
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; Initial or prolonged in-patient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug to the end of study (up to Day 30) that were absent before treatment or that worsened relative to pre-treatment state. AEs included both serious and non-serious adverse events.
Time Frame: Baseline (Day 1) up to Day 30
Population: Safety analysis set included all participants who received at least 1 dose of study medication (L-Dopa or PF-06649751) in Period 1 and/or Period 2.
Measure: Number; unit: participants
Arm/Group | L-Dopa | PF-06649751 5 mg + L-Dopa | PF-06649751 15 mg + L-Dopa | PF-06649751 15 mg + L-Dopa: L-dopa Induced Dyskinesia (LID) | PF-06649751 25 mg + L-Dopa
Number analyzed (Participants) | 50 | 9 | 11 | 6 | 19
participants
  AEs | 9 | 9 | 7 | 5 | 15
  SAEs | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Criteria for laboratory abnormalities: Hemoglobin (Hgb),hematocrit, red blood cell(RBC) count: less than(<)0.8*lower limit of normal(LLN),mean corpuscular Hgb, mean corpuscular volume, mean corpuscular Hgb concentration:<0.9*LLN, greater than (>)1.1*upper limit of normal(ULN),platelet:<0.5*LLN,>1.75*ULN,lymphocyte,neutrophil:<0.8*LLN, >1.2*ULN, basophil, eosinophil, monocyte:>1.2*ULN, WBC:<0.6*LLN, >1.5*ULN;total bilirubin>1.5*ULN, aspartate aminotransferase,alanine aminotransferase,alkaline phosphatase:>3.0*ULN,total protein,albumin:<0.8*LLN,>1.2*ULN;blood urea nitrogen,creatinine:>1.3*ULN, uric acid>1.2*ULN;sodium<0.95*LLN,>1.05*ULN,potassium,chloride,calcium,bicarbonate:<0.9*LLN,>1.1*ULN;glucose<0.6*LLN,>1.5*ULN,urine pH:<4.5, >8; urine: WBC, RBC greater than or equal to (>=)20/high performance field, bacteria: >20; urobilinogen, urine: glucose, ketone, protein, Hgb, nitrite, leukocyte esterase, bilirubin: >=1.
Time Frame: Baseline up to Day 30
Population: Safety analysis set included all participants who received at least 1 dose of study medication (L-Dopa or PF-06649751) in Period 1 and/or Period 2. Here, number of participants analyzed (N) signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | L-Dopa | PF-06649751 5 mg + L-Dopa | PF-06649751 15 mg + L-Dopa | PF-06649751 15 mg + L-Dopa: L-dopa Induced Dyskinesia (LID) | PF-06649751 25 mg + L-Dopa
Number analyzed (Participants) | 49 | 9 | 11 | 6 | 18
participants | 17 | 8 | 8 | 5 | 11

3. Primary Outcome: Number of Participants With Vital Sign Abnormalities
Description: Criteria for vital sign abnormality included supine pulse rate of <40 beats per minute (bpm) or >120 bpm, standing pulse rate of <40 bpm or >140 bpm, supine and standing systolic blood pressure (SBP) <90 millimeter of mercury (mmHg), supine and standing diastolic blood pressure (DBP) <50 mmHg, supine and standing SBP of >=30 mmHg maximum (max.) increase from baseline (IFB) and and decrease from baseline (DFB) in same posture, supine and Standing DBP of >=20 mmHg max. increase and decrease from baseline in same posture. Categories in which there was atleast 1 abnormality are reported in this outcome measure.
Time Frame: Baseline up to Day 30
Population: Safety analysis set included all participants who received at least 1 dose of study medication (L-Dopa or PF-06649751) in Period 1 and/or Period 2. Here, 'n' signifies the number of participants evaluable for the specific category.
Measure: Number; unit: participants
Arm/Group | L-Dopa | PF-06649751 5 mg + L-Dopa | PF-06649751 15 mg + L-Dopa | PF-06649751 15 mg + L-Dopa: L-dopa Induced Dyskinesia (LID) | PF-06649751 25 mg + L-Dopa
Number analyzed (Participants) | 50 | 9 | 11 | 6 | 19
participants
  Supine SBP: <90 mmHg (n =50, 9, 11, 6, 19) | 2 | 1 | 1 | 1 | 1
  Standing SBP: <90 mmHg (n =50, 9, 11, 6, 19) | 5 | 2 | 3 | 1 | 0
  Supine DBP: <50 mmHg (n =50, 9, 11, 6, 19) | 1 | 1 | 0 | 0 | 1
  Max. IFB in Supine SBP: >=30 mmHg (n=50,9,11,6,19) | 1 | 2 | 1 | 0 | 2
  Max. IFB in StandingSBP:>=30 mmHg(n= 49,9,11,6,19) | 3 | 1 | 0 | 0 | 2
  Max. IFB in Supine DBP: >=20 mmHg(n= 50,9,11,6,19) | 1 | 1 | 2 | 0 | 1
  Max. IFB in StandingDBP:>=20 mmHg(n= 49,9,11,6,19) | 1 | 0 | 0 | 0 | 2
  Max. DFB in Supine SBP:>=30 mmHg (n= 50,9,11,6,19) | 8 | 1 | 3 | 1 | 5
  Max. DFB in StandingSBP:>=30 mmHg(n= 49,9,11,6,19) | 7 | 2 | 4 | 2 | 4
  Max. DFB in Supine DBP:>=20 mmHg (n= 50,9,11,6,19) | 9 | 3 | 2 | 3 | 8
  Max. DFB in StandingDBP:>=20 mmHg(n= 49,9,11,6,19) | 11 | 2 | 3 | 2 | 5

4. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: Criteria for ECG abnormalities: maximum PR interval >=300 milliseconds (msec) and maximum increase PR interval increase from baseline (IFB): percent change (Pctchg) >=25 percent (%) for baseline value of >200 msec and Pctchg>=50% for baseline value of <=200 msec for PR interval, maximum QRS interval >=140 msec and a maximum IFB: Pctchg>=50%, maximum QTCF interval (Fridericia's Correction) of 450 msec to <480 msec, 480 msec to <500 msec or >=500 msec and a maximum change of <=30change<60 or >=60 msec from baseline.
Time Frame: Baseline up to Day 30
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | L-Dopa | PF-06649751 5 mg + L-Dopa | PF-06649751 15 mg + L-Dopa | PF-06649751 15 mg + L-Dopa: L-dopa Induced Dyskinesia (LID) | PF-06649751 25 mg + L-Dopa
Number analyzed (Participants) | 50 | 9 | 11 | 5 | 18
participants | 2 | 0 | 2 | 1 | 2

5. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Physical Examination Findings
Description: Physical examination included examination of the head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems. The examination assessed the participants for any potential changes in general appearance, the respiratory and cardiovascular systems, as well as towards participant reported symptoms. Findings were considered to be clinically significant based on investigator's decision.
Time Frame: Baseline up to Day 30
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | L-Dopa | PF-06649751 5 mg + L-Dopa | PF-06649751 15 mg + L-Dopa | PF-06649751 15 mg + L-Dopa: L-dopa Induced Dyskinesia (LID) | PF-06649751 25 mg + L-Dopa
Number analyzed (Participants) | 50 | 9 | 11 | 6 | 19
participants | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Clinically Significant Neurological Examination Abnormality
Description: The complete or full neurological examination included assessment of the cranial nerves; muscle strength, tone, cortical drift, abnormal movements; deep tendon reflexes; sensory exam, coordination, gait and station. Higher cortical and motor function was considered part of the complete neurological exam. Findings were considered abnormal as confirmed by a certified neurologist.
Time Frame: Baseline up to Day 30
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | L-Dopa | PF-06649751 5 mg + L-Dopa | PF-06649751 15 mg + L-Dopa | PF-06649751 15 mg + L-Dopa: L-dopa Induced Dyskinesia (LID) | PF-06649751 25 mg + L-Dopa
Number analyzed (Participants) | 50 | 9 | 11 | 6 | 19
participants | 0 | 0 | 0 | 0 | 1

7. Primary Outcome: Number of Participants With Categorical Scores on The Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS was an interview-based rating scale to systematically assess suicidal ideation and suicidal behavior. C-SSRS assessed whether participant experienced any of the following 1: completed suicide, 2: suicide attempt (response of "yes" on "actual attempt"), 3: preparatory acts toward imminent suicidal behavior ("yes" on "aborted attempt", "interrupted attempt", "preparatory acts or behavior"), 4: any suicidal behavior or ideation, suicidal ideation ("yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent"), 7: self-injurious behavior, no suicidal intent ("yes" on "has participant engaged in non-suicidal self-injurious behavior").
Time Frame: Baseline up to Day 30
Population: Safety analysis set included all participants who received at least 1 dose of study medication (L-Dopa or PF-06649751) in Period 2. This outcome measure was not planned to be assessed in lead-in period (L-dopa).
Measure: Number; unit: participants
Arm/Group | PF-06649751 5 mg + L-Dopa | PF-06649751 15 mg + L-Dopa | PF-06649751 15 mg + L-Dopa: L-dopa Induced Dyskinesia (LID) | PF-06649751 25 mg + L-Dopa
Number analyzed (Participants) | 9 | 11 | 6 | 19
participants | 0 | 0 | 0 | 0

8. Primary Outcome: Change From Baseline in Parkinson's Disease Diary For Participants With Motor Fluctuations at Day 13
Description: According to Parkinson's disease diaries of participants "OFF" time was a time period when the medication no longer providing benefit with regard to mobility, slowness, and stiffness and participants experienced relatively poor overall function with worsening of tremor, rigidity, balance, or bradykinesia. "ON" time was a time period when medication was providing benefit with regard to mobility, slowness, and stiffness. "ON" time was classified as associated with or without troublesome dyskinesia (TD) that interfere with activities of daily living and with or without dyskinesia. "OFF" time and "ON" time with TD were generally considered to be "bad time" with regard to motor function, whereas "ON" time without dyskinesia (WD) and with non- troublesome dyskinesia (NTD) were generally considered to be "good time".
Time Frame: Baseline, Day 13
Population: Safety analysis set included all participants who received at least 1 dose of study medication(L-Dopa or PF-06649751) in Period 2. Here,'n' signifies those participants who were evaluable at specified time points for each reporting arm.This outcome measure was not planned to be assessed in lead-in period (L-dopa).
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | PF-06649751 5 mg + L-Dopa | PF-06649751 15 mg + L-Dopa | PF-06649751 15 mg + L-Dopa: L-dopa Induced Dyskinesia (LID) | PF-06649751 25 mg + L-Dopa
Number analyzed (Participants) | 9 | 11 | 6 | 19
hour
  Total OFF time: Baseline (n=9,11,6,19) | 4.42 (5.073) | 6.18 (3.433) | 6.75 (1.789) | 6.05 (3.981)
  Total OFF time: Change at Day 13 (n=9,9,3,9) | -0.14 (3.310) | -0.31 (4.976) | 1.75 (2.646) | -2.44 (6.335)
  Total ON time: Baseline (n=9,11,6,19) | 11.92 (5.328) | 9.52 (3.665) | 8.13 (3.485) | 10.96 (4.862)
  Total ON time: Change at Day 13 (n=9,9,3,9) | 1.86 (4.150) | 1.81 (6.644) | -4.25 (0.750) | 0.06 (6.232)
  ON time WD: Baseline (n=9, 11, 6, 19) | 7.58 (5.995) | 8.59 (2.996) | 4.13 (3.781) | 9.14 (5.950)
  ON time WD: Change at Day 13 (n=9, 9, 3, 9) | -1.50 (4.081) | 1.86 (6.519) | -1.75 (3.031) | -0.78 (4.604)
  ON time with dyskinesia: Baseline (n=9,11,6,19) | 4.33 (5.851) | 0.93 (1.946) | 4.00 (3.698) | 1.82 (3.326)
  ON time with dyskinesia:Change at Day13(n=9,9,3,9) | 3.36 (5.460) | -0.06 (0.891) | -2.50 (2.411) | 0.83 (6.294)
  ON time with TD: Baseline (n=9, 11, 6, 19) | 1.56 (2.518) | 0.36 (0.876) | 0.29 (0.510) | 0.43 (1.833)
  ON time with TD: Change at Day 13 (n=9, 9, 3, 9) | 1.58 (2.469) | -0.14 (0.417) | 0.25 (0.433) | -0.67 (2.000)
  Good ON time: Baseline (n=9, 11, 6, 19) | 10.36 (5.053) | 9.16 (3.181) | 7.83 (3.319) | 10.53 (5.165)
  Good ON time: Change at Day 13 (n=9, 9, 3, 9) | 0.28 (2.830) | 1.94 (6.690) | -4.50 (1.146) | 0.72 (5.906)
  Total Awake time: Baseline (n=9, 11, 6, 19) | 16.33 (1.620) | 15.70 (1.495) | 14.88 (2.602) | 17.01 (4.063)
  Total Awake time: Change at Day 13 (n=9, 9, 3, 9) | 1.72 (1.748) | 1.50 (3.267) | -2.50 (2.883) | -2.39 (5.456)
  Total Asleep time: Baseline (n=9, 11, 6, 19) | 7.67 (1.620) | 8.30 (1.495) | 7.92 (2.053) | 6.24 (2.895)
  Total Asleep time: Change at Day 13 (n=9, 9, 3, 9) | -1.72 (1.748) | -1.50 (3.267) | -0.33 (2.626) | 0.44 (0.982)

9. Primary Outcome: Change From Baseline in Parkinson's Disease Diary For Participants With Motor Fluctuations at Day 20
Description: as for outcome 8
Time Frame: Baseline, Day 20
Population: Safety analysis set included all participants who received at least 1 dose of study medication(L-Dopa or PF-06649751) in Period 2. Here,'n' signifies those participants who were evaluable at specified time points for each reporting arm. This outcome measure was not planned to be assessed in lead-in period (L-dopa).
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | PF-06649751 5 mg + L-Dopa | PF-06649751 15 mg + L-Dopa | PF-06649751 15 mg + L-Dopa: L-dopa Induced Dyskinesia (LID) | PF-06649751 25 mg + L-Dopa
Number analyzed (Participants) | 9 | 9 | 2 | 8
hour
  Total OFF time: Change at Day 20 | 1.97 (3.166) | -0.19 (2.965) | 0.63 (4.419) | -1.94 (5.603)
  Total ON time: Change at Day 20 | -1.53 (3.556) | 0.69 (3.739) | -0.63 (3.005) | 0.66 (6.518)
  ON time WD: Change at Day 20 | -2.61 (3.814) | 1.06 (3.980) | -2.13 (3.005) | -0.41 (3.659)
  ON time with dyskinesia: Change at Day 20 | 1.08 (5.297) | -0.36 (0.730) | 1.50 (6.010) | 1.06 (8.174)
  ON time with TD: Change at Day 20 | 0.47 (1.910) | -0.08 (0.468) | 0.25 (0.000) | -0.66 (1.856)
  Good ON time: Change at Day 20 | -2.00 (2.613) | 0.78 (3.768) | -0.88 (3.005) | 1.31 (6.088)
  Total Awake time: Change at Day 20 | 0.44 (1.116) | 0.50 (2.154) | 0.00 (1.414) | -1.28 (1.538)
  Total Asleep time: Change at Day 20 | -0.44 (1.116) | -0.50 (2.154) | 0.00 (1.414) | 1.28 (1.538)

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of L-Dopa
Time Frame: Pre-dose, 0.5, 1, 2, 4 and 8 hours post-dose on Day 1
Population: The L-Dopa pharmacokinetic (PK) parameter analysis set included all participants who received at least 1 dose of L-Dopa in open label Period 1 with at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | L-Dopa
Number analyzed (Participants) | 50
nanogram per milliliter (ng/mL) | 2817 (60)

11. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of L-Dopa
Time Frame: Pre-dose, 0.5, 1, 2, 4 and 8 hours post-dose on Day 1
Population: The L-Dopa PK parameter analysis set included all participants who received at least 1 dose of L-Dopa in open label Period 1 with at least 1 of the PK parameters of interest.
Measure: Median (Full Range); unit: hour
Arm/Group | L-Dopa
Number analyzed (Participants) | 50
hour | 0.517 [0.417 to 8.25]

12. Secondary Outcome: Apparent Clearance (CL/F) of L-Dopa
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Pre-dose, 0.5, 1, 2, 4 and 8 hours post-dose on Day 1
Population: The L-Dopa PK parameter analysis set included all participants who received at least 1 dose of L-Dopa in open label Period 1 with at least 1 of the PK parameters of interest. Here, number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/hr)
Arm/Group | L-Dopa
Number analyzed (Participants) | 42
liter per hour (L/hr) | 33.57 (37)

13. Secondary Outcome: Terminal Half-Life (t1/2) of L-Dopa
Description: Terminal half-life is the time measured for the plasma concentration of drug to decrease by one half. It was calculated as dividing the natural logarithm to the base e (Log e)*2/k el, where k el is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Pre-dose, 0.5, 1, 2, 4 and 8 hours post-dose on Day 1
Population: The L-Dopa PK parameter analysis set included all participants who received at least 1 dose of L-Dopa in open label Period 1 with at least 1 of the PK parameters of interest. Here, number of participants analyzed (N) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | L-Dopa
Number analyzed (Participants) | 42
hour | 1.534 (0.23847)

14. Secondary Outcome: Area Under the Curve From Time Zero Extrapolated to Infinite Time of L-Dopa
Description: AUC (0 - inf)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - inf). It is obtained from AUC (0 - t) plus AUC (t - inf).
Time Frame: Pre-dose, 0.5, 1, 2, 4 and 8 hours post-dose on Day 1
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | L-Dopa
Number analyzed (Participants) | 42
nanogram*hour per milliliter (ng*hr/mL) | 6117 (57)

15. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration of L-Dopa
Description: Area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration (C last).
Time Frame: Pre-dose, 0.5, 1, 2, 4 and 8 hours post-dose on Day 1
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | L-Dopa
Number analyzed (Participants) | 50
ng*hr/mL | 6152 (56)

16. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of L-Dopa
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: Pre-dose, 0.5, 1, 2, 4 and 8 hours post-dose on Day 1
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | L-Dopa
Number analyzed (Participants) | 42
Liter (L) | 73.41 (41)

17. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-06649751
Time Frame: Pre-dose on Day 3, 4, 8, 11, 14, 17, 20, Pre-dose, 0.5, 1, 1.5, 2, 4, 8 and 12 hour post-dose on Day 7, 13, 22
Population: The PF-06649751 PK parameter analysis set included all participants treated and who had at least 1 of the PK parameters of interest in at least 1 treatment period during period 2. Here, 'n' signifies those participants who were evaluable at specified time points for each reporting arm, respectively.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06649751 5 mg + L-Dopa | PF-06649751 15 mg + L-Dopa | PF-06649751 15 mg + L-Dopa: L-dopa Induced Dyskinesia (LID) | PF-06649751 25 mg + L-Dopa
Number analyzed (Participants) | 9 | 11 | 6 | 19
ng/mL
  Day 7 (n =9, 9, 5, 14) | 18.95 (51) | 53.69 (41) | 31.72 (25) | 68.17 (23)
  Day 13 (n =9, 7, 3, 5) | 79.87 (27) | 215.7 (48) | 143.6 (27) | 309.0 (20)
  Day 22 (n =9, 7, 3, 7) | 118.5 (33) | 325.4 (46) | 241.2 (26) | 401.6 (41)

18. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-06649751
Time Frame: Pre-dose on Day 3, 4, 8, 11, 14, 17, 20, Pre-dose, 0.5, 1, 1.5, 2, 4, 8 and 12 hour post-dose on Day 7, 13, 22
Population: The PF-06649751 PK parameter analysis set included all participants treated and who had at least 1 of the PK parameters of interest in at least 1 treatment period during period 2. Here, 'n' signifies those participants who were evaluable at specified time point for each reprting arm, respectively.
Measure: Median (Full Range); unit: hour
Arm/Group | PF-06649751 5 mg + L-Dopa | PF-06649751 15 mg + L-Dopa | PF-06649751 15 mg + L-Dopa: L-dopa Induced Dyskinesia (LID) | PF-06649751 25 mg + L-Dopa
Number analyzed (Participants) | 9 | 11 | 6 | 19
hour
  Day 7 (n =9, 9, 5, 14) | 1.00 [0.500 to 4.00] | 2.45 [1.03 to 4.15] | 2.00 [1.75 to 4.00] | 3.18 [0.500 to 11.6]
  Day 13 (n =9, 7, 3, 1) | 2.00 [0.833 to 12.0] | 3.92 [2.03 to 11.8] | 2.00 [2.00 to 4.00] | 8.00 [8.00 to 8.00]
  Day 22 (n =9, 7, 3, 7) | 2.00 [1.00 to 4.00] | 4.00 [2.00 to 12.0] | 2.02 [2.00 to 4.00] | 4.03 [1.97 to 8.00]

19. Secondary Outcome: Apparent Clearance (CL/F) of PF-06649751
Description: as for outcome 12
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 4, 8 and 12 hour post-dose on Day 22
Population: The PF-06649751 PK parameter analysis set included all participants treated and who had at least 1 of the PK parameters of interest in at least 1 treatment period during period 2. Here, number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | PF-06649751 5 mg + L-Dopa | PF-06649751 15 mg + L-Dopa | PF-06649751 15 mg + L-Dopa: L-dopa Induced Dyskinesia (LID) | PF-06649751 25 mg + L-Dopa
Number analyzed (Participants) | 9 | 7 | 3 | 7
L/hr | 2.377 (35) | 2.504 (61) | 3.511 (40) | 3.483 (52)

20. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval of PF-06649751
Description: Area under the concentration curve from time zero to end of dosing interval (AUCtau), where dosing interval was 12 hours.
Time Frame: Pre-dose on Day 3, 4, 8, 11, 14, 17, 20, Pre-dose, 0.5, 1, 1.5, 2, 4, 8 and 12 hour post-dose on Day 7, 13, 22
Population: The PF-06649751 PK parameter analysis set included all participants treated and who had at least 1 of the PK parameters of interest in at least 1 treatment period during period 2. Here, 'n' signifies those participants who were evaluable at specified time point for each reporting arm, respectively.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06649751 5 mg + L-Dopa | PF-06649751 15 mg + L-Dopa | PF-06649751 15 mg + L-Dopa: L-dopa Induced Dyskinesia (LID) | PF-06649751 25 mg + L-Dopa
Number analyzed (Participants) | 9 | 11 | 6 | 19
ng*hr/mL
  Day 7 (n =9, 9, 5, 14) | 261.9 (30) | 990.8 (56) | 530.9 (30) | 1203 (25)
  Day 13 (n =9, 7, 3, 5) | 1438 (30) | 4192 (61) | 2414 (39) | 5498 (32)
  Day 22 (n =9, 7, 3, 7) | 2105 (35) | 5993 (61) | 4271 (40) | 7182 (52)

21. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) of PF-06649751
Time Frame: Pre-dose on Day 3, 4, 8, 11, 14, 17, 20, Pre-dose, 0.5, 1, 1.5, 2, 4, 8 and 12 hour post-dose on Day 7, 13, 22
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06649751 5 mg + L-Dopa | PF-06649751 15 mg + L-Dopa | PF-06649751 15 mg + L-Dopa: L-dopa Induced Dyskinesia (LID) | PF-06649751 25 mg + L-Dopa
Number analyzed (Participants) | 9 | 11 | 6 | 19
ng/mL
  Day 7 (n =9, 9, 5, 14) | 7.295 (30) | 27.97 (66) | 14.19 (38) | 24.29 (36)
  Day 13 (n =9, 7, 3, 5) | 35.00 (69) | 132.5 (77) | 65.19 (56) | 162.3 (37)
  Day 22 (n =9, 7, 3, 7) | 68.14 (44) | 197.9 (78) | 120.8 (68) | 215.1 (63)

22. Secondary Outcome: Ratio of Accumulation for Area Under the Curve From Time Zero to End of Dosing Interval of PF-06649751
Description: Rac was obtained from AUCtau after last dose divided by AUCtau after first dose, where AUC(tau) = Area under the concentration curve from time zero to end of dosing interval (AUCtau), where dosing interval was 12 hours.
Time Frame: Pre-dose on Day 3, 4, 8, 11, 14, 17, 20, Pre-dose, 0.5, 1, 1.5, 2, 4, 8 and 12 hour post-dose on Day 7, 13, 22
Population: Data was not collected since this outcome measure was not planned to be analyzed.
Arm/Group | PF-06649751 5 mg + L-Dopa | PF-06649751 15 mg + L-Dopa | PF-06649751 15 mg + L-Dopa: L-dopa Induced Dyskinesia (LID) | PF-06649751 25 mg + L-Dopa
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to Day 30
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | L-Dopa | PF-06649751 5 mg + L-Dopa | PF-06649751 15 mg + L-Dopa | PF-06649751 15 mg + L-Dopa: L-dopa Induced Dyskinesia (LID) | PF-06649751 25 mg + L-Dopa
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/9 | 0/11 | 0/6 | 1/19
Other Adverse Events (participants affected / at risk) | 8/50 | 9/9 | 7/11 | 5/6 | 15/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | L-Dopa (N=50) | PF-06649751 5 mg + L-Dopa (N=9) | PF-06649751 15 mg + L-Dopa (N=11) | PF-06649751 15 mg + L-Dopa: L-dopa Induced Dyskinesia (LID) (N=6) | PF-06649751 25 mg + L-Dopa (N=19)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | L-Dopa (N=50) | PF-06649751 5 mg + L-Dopa (N=9) | PF-06649751 15 mg + L-Dopa (N=11) | PF-06649751 15 mg + L-Dopa: L-dopa Induced Dyskinesia (LID) (N=6) | PF-06649751 25 mg + L-Dopa (N=19)
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Blepharospasm (Eye disorders) | 0 | 1 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 0 | 3 | 2 | 8
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 4
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1
Drug withdrawal syndrome (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 0 | 1 | 0
Infusion site swelling (General disorders) | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Posture abnormal (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 2 | 5
Dystonia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Freezing phenomenon (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 6 | 7 | 3 | 8
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 2 | 0 | 2 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 3 | 2 | 1 | 3
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 2 | 1
Depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Dysphoria (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Hallucination, auditory (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 3 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 1 | 1 | 0 | 2 | 2
Sleep terror (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.